CLINICAL TRIAL: NCT05954364
Title: Sex Matters: Sex- And Gender-based Analysis of the Effectiveness of Advanced Therapies in Psoriatic Arthritis (SAGE-PsA) - an International Multicentre Study
Brief Title: Sex and Gender-based Analysis of the Effectiveness of Advanced Therapies in Psoriatic Arthritis
Acronym: SAGE-PsA
Status: Recruiting | Type: Observational
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Lihi Eder, Associate Professor, Department of Medicine, University of Toronto
Other Study IDs: 2022-0095-B
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Inflammatory Arthritis; Sex; Gender; Advanced Therapies
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be collected in selected sites that have a capacity to collect, process and store these samples locally prior to shipment to the coordinating site. These samples will be collected during the baseline and follow-up in person visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic Arthritis: Patients with a rheumatologist-confirmed diagnosis of psoriatic arthritis who are initiating advanced therapy for peripheral musculoskeletal manifestations of psoriatic arthritis

SUMMARY:
Sex and gender are important factors that influence treatment response in PsA. The goal of this multi-centre observational study is to understand how sex and gender influence response to advanced therapies in psoriatic arthritis (PsA). The investigators hope to discover biological and socio-cultural mechanisms that explain the differences in treatment response between men and women with PsA.

The study investigators plan to recruit patients from approximately 30 sites across the world. Men and women with active PsA will be assessed before and after they start advanced therapies and information will be collected about sex- and gender-related factors through questionnaires and physical examination. Physicians will assess the patient response to treatment. The investigators will compare the response to treatment in men and women and assess what biological and socio-cultural factors contribute to differences in treatment response.

DETAILED DESCRIPTION:
Study investigators will perform a prospective, multi-center, international cohort study involving approximately 30 sites that specialize in care of patients with PsA. 540 patients with a rheumatologist-confirmed diagnosis of PsA who are initiating advanced therapy for peripheral musculoskeletal manifestations of PsA will be enrolled. The study will include 2 in-person physician visits. Visit 1 (baseline) will take place prior to drug initiation (up to 3 months prior). Visit 2 (follow-up) will occur 3-6 months following drug initiation. In addition, study sites will be asked to report persistence status on the study drug at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologist confirmed diagnosis of PsA according to CASPAR criteria
* Age ≥18 years
* Active PsA with any of the following manifestations detected on physical examination: peripheral arthritis, dactylitis, and enthesitis. The patient may have axial involvement in addition to the peripheral manifestations of PsA
* Plan to start treatment with advanced therapies for peripheral musculoskeletal manifestations of PsA

Exclusion Criteria:

* Unable to read or write
* Unable to sign informed consent
* Cannot return for a follow up visit
* The drug is given for another indication and not for active PsA (e.g. psoriasis, IBD)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients with psoriatic arthritis who have been identified in clinic by their rheumatologist
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of the American College of Rheumatology (ACR) 20/50/70 | Within 3-6 months
  The proportion of patients who have achieved the ACR 20/50/70 following treatment initiation
Achievement of Minimal Disease Activity (MDA) state | Within 3-6 months
  The proportion of patients who have achieved the MDA state following treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Lihi Eder, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided